CLINICAL TRIAL: NCT05184738
Title: Evaluation of the Tolerance of Two Oral Nutritional Supplements in Patients with Anorexia Nervosa
Brief Title: Nutritional Supplements in Patients with Anorexia Nervosa
Acronym: PEPTIDICAN21
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PEPTIDIC-AN-2021
Record Dates: First submitted 2021-12-02; First posted 2022-01-11 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia nervosa; malnutrition; oligomeric formula; polymeric formula; digestive tolerance; body composition; functional capacity; quality of life; anxiety; depression
MeSH Terms: conditions — Anorexia Nervosa; Malnutrition; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oligomeric nutritional formula arm (Bi1 peptidic) (Experimental): Individuals will receive a Oligomeric nutritional formula.
  Interventions: Other: Experimental Treatment, Oligomeric nutritional formula
- Standard arm (Other): Individuals will receive a Standard nutritional formula.
  Interventions: Other: Control Treatment

INTERVENTIONS:
Other: Experimental Treatment, Oligomeric nutritional formula — Intervention group will receive a oligomeric nutritional formula (Bi1 peptidic Adventia Pharma, Spain).
  Arms: Oligomeric nutritional formula arm (Bi1 peptidic)
Other: Control Treatment — Standard nutritional formula (isocaloric and isoprotein compared to the experimental treatment).
  Arms: Standard arm

SUMMARY:
Anorexia nervosa causes gastroparesis, constipation, and can lead to elevated liver enzymes. It is often necessary to supplement the diet of patients with nutritional formulas. The ingestion of a peptide formula, with partially hydrolyzed protein and rich in medium chain triglycerides, could favor its digestion and absorption, improving its tolerance and acceptance by the patient, compared to a polymeric formula.

DETAILED DESCRIPTION:
Main objective:

• To compare the digestive tolerance of an oligomeric nutritional supplement with respect to a polymeric nutritional supplement in a group of patients diagnosed with anorexia nervosa under follow-up by the Nutrition Unit.

Secondary Objectives:

* Assess the gastrointestinal tolerance of the oral nutritional supplement on a single occasion with respect to a continuous intake over a period of 4 weeks.
* Evaluate the impact of oral nutritional supplementation on nutritional status over a four-week period.
* Evaluate the impact of oral nutritional supplementation on the functional capacity of the patient in a period of four weeks.
* Evaluate the impact of oral nutritional supplementation on the patient's body composition over a four-week period.
* Evaluate the impact of oral nutritional supplementation on the quality of life of the patient in a period of four weeks.
* Evaluate the impact of oral nutritional supplementation on the depressive and anxious symptoms of the patient in a period of four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, ≥ 12 y ≤ 40 years of age at screening
* Diagnosed of Anorexy nervous according to DSM-5
* Appropiate cultural level & understanding of the clinical study
* To be in agreement in participate voluntarily in the study and written informed consent must be obtained from the participants.
* Females who are non-pregnant and non-lactating women or women who have given birth at least six weeks before to the screening visit.

Exclusion Criteria:

* Allergy or intolerance to any component of the products under study.
* Participation in a concomitant trial that conflicts with this study
* Doesn't sign the informed consent

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-03-12 (Actual); Study Completion 2022-05-22 (Actual)

PRIMARY OUTCOMES:
Compare the digestive tolerance of an oligomeric nutritional supplement with respect to a polymeric nutritional supplement in a group of patients diagnosed with anorexia nervosa under follow-up by the Nutrition Unit. | From baseline to week 1
  Differences in the score of the questionnaire: "Evaluation questionnaire for gastrointestinal complaints". This questionnaire assesses the presence (and where appropriate its degree) or absence of nausea, vomiting, diarrhea, constipation, reflux or heartburn. Each section has a score from 0 to 10, which will be filled in by the patient himself.

SECONDARY OUTCOMES:
Assess the gastrointestinal tolerance of the oral nutritional supplement on a single occasion with respect to a continuous intake over a period of 4 weeks. | From baseline to week 1 in group 1; from baseline to week 8 in group 2
  Difference in score in the questionnaire "Evaluation questionnaire for gastrointestinal complaints". This questionnaire assesses the presence (and where appropriate its degree) or absence of nausea, vomiting, diarrhea, constipation, reflux or heartburn. Each section has a score from 0 to 10, which will be filled in by the patient himself.
Compare the sensory perception of a polymeric nutritional supplement with respect to an oligomeric one. | From baseline to week 1 in group 1; from baseline to week 8 in group 2
  Change in the score of the "Product sensory evaluation questionnaire". It consists of 11 items, which assess how the patient perceives the organoleptic characteristics of the product and their satisfaction after taking it. Each item consists of a score from 0 to 10 that the patient has to fill in. The items can refer to positive or negative characteristics of the product, so the level of score in each of them can indicate better or worse characteristics of the product depending on the characteristic in question.
Compare adherence to treatment in group 2 subjects. | From baseline to week 8 in group 2
  Adherence will be determined by daily registration of the percentage they take of the supplement.
Evaluate the intake of natural food in group 2 patients. | From baseline to week 8 in group 2
  Dietary registration of natural food intake at breakfast, mid-morning snack and lunch, in group 2 patients. It will be done through the DIETSTAT program. The total amount of calories and the percentage of macronutrients will be determined.
Changes in weight | From baseline to week 8
  Weight will be measured in kg
Change in hand grip strength | From baselilne to week 8
  It will be determined with a JAMAR dynamometer. The mean and maximum of three measurements made on the dominant hand and the mean and maximum of three measurements made on the non-dominant hand will be taken. The outside will be measured in kg.
Change in fat mass | From baselilne to week 8
  Determined by AKERN bioimpedance analyzer and measured in kg
Change in lean mass | From baselilne to week 8
  Determined by AKERN bioimpedance meter and measured in kg
Change in extracellular water | From baselilne to week 8
  Determined by AKERN bioimpedance analyzer and measured in l
Change in intracellular water | From baselilne to week 8
  Determined by AKERN bioimpedance analyzer and measured in l
Change in phase angle | From baselilne to week 8
  Determined by AKERN bioimpedance analyzer and measured in degrees of angle
Change in total cell mass | From baselilne to week 8
  Determined by AKERN bioimpedance analyzer and measured in kg
Evaluate the impact of oral nutritional supplementation on the quality of life of the patient | From baselilne to week 8
  Changes in the score of the "SF-12 Health Questionnaire" questionnaire. This questionnaire is the adaptation made for Spain of the SF-12 Health Survey. The SF-12 is a shortened version of the SF-36 Health Questionnaire designed for uses where it is too long. Provides a health status profile. It consists of 12 items from the 8 dimensions of the SF-36 Physical Function (2), Social Function (1), Physical role (2), Emotional role (2), Mental health (2), Vitality (1), Body pain (1), General Health (1). The response options form Likert-type scales that assess intensity or frequency. The number of answer options ranges from three to six, depending on the item. For each of the 8 dimensions, the items are coded, added and transformed on a scale that ranges from 0 (the worst health status for that dimension) to 100 (the best health status).
Changes in eating habits and styles | From baselilne to week 8
  Changes in the score of the "Eating Disorder Examination-Q (EDE-Q)" test. This questionnaire takes about 10 minutes to complete. It studies the scope and severity of the characteristics associated with the diagnosis of eating disorder. It includes 4 subscales: Restriction-diet, Preoccupation with food, Preoccupation with weight and Concern about the figure. Includes a definition of the term "binge" (eg, "episodes in which you have eaten an abnormally large amount of food under the circumstances" and experiencing a "loss of control" over eating). The EDE-Q generates two types of data: frequency data on key behavioral features of eating disorders in terms of number of episodes of the behavior, and subscale scores reflecting the severity of characteristics of eating disorders. Higher scores on the global scale and subscales denote more problematic eating behaviors and attitudes.
Assess the impact of oral nutritional supplementation on the patient's depressive and anxious symptoms. | From baseline to week 8
  Changes in the score of the "Hospital Anxiety and Depression Scale (HADS)". This aims to detect depressive and anxiety disorders in non-psychiatric hospital services, avoiding overlap with symptoms due to physical illness, without taking into account the physical aspects that may accompany anxiety / depression, only affecting the emotional ones. It is a self-administered scale with 14 items divided into 2 subscales (anxiety and depression) whose maximum score is 21 points for each of them. Based on the score obtained, patients can be classified as normal (<7), doubtful (between 8 and 10) and potential clinical case (≥ 11). The score is referred to the last week.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel MD Olveira, PhD, Principal Investigator — Hospital Regional Universitario de Málaga, FIMABIS
Locations (1):
- Hospital Regional Universitario de Málaga, Málaga, MALAGA, Spain

REFERENCES:
- [Derived] Ruiz Garcia I, Porras Perez N, Garcia Torres F, Olivas Delgado L, Sanchez Torralvo FJ, Pascual Lopez M, Fernandez Marzalo C, Olveira G. Comparison of the digestive tolerance of an oligomeric versus a polymeric oral nutritional supplement in people with anorexia nervosa. A randomised crossover clinical trial. Eur J Clin Nutr. 2025 Aug;79(8):780-786. doi: 10.1038/s41430-025-01608-y. Epub 2025 Mar 31. PMID 40164776